CLINICAL TRIAL: NCT02368457
Title: Advances in the Management of Mandibular Osteoradionecrosis: Pentoxifylline and Tocopherol as Medical Treatment
Brief Title: Management of Mandibular ORN: PENTO as Medical Treatment
Acronym: PENTO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Miriam Martos-Fernandez, Oral and Maxillofacial Surgeon, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORN-2014-16
Record Dates: First submitted 2015-02-10; First posted 2015-02-23 (Estimated); Results first posted 2016-12-20 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Osteoradionecrosis
Keywords: Mandibular osteoradionecrosis; Tocopherol; pentoxifylline; vitamine E; wounds and injuries; antioxidants; free radical scavengers; radiation-protective agents; vasodilatadors agents; osteonecrosis; mandible; extraoral fistula; exposed bone; necrotic bone; head and neck radiotherapy
MeSH Terms: conditions — Osteoradionecrosis; Wounds and Injuries; Osteonecrosis | interventions — Pentoxifylline; Tocopherols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pentoxifylline and Tocopherol (Experimental): Drug: pentoxifylline with tocopherol Combination of pentoxifylline and tocopherol during a minimum of 6 months and a maximum of 24 months.
  Interventions: Drug: Pentoxifylline and Tocopherol
- CONTROL (No Intervention): No drug treatment

INTERVENTIONS:
Drug: Pentoxifylline and Tocopherol — pentoxifylline with tocopherol Pentoxifylline 800 mg/day, oral (1cp 400 mg twice a day) + Vitamin E (alfa-tocopherol) 1000 UI/day, oral (1cp 400UI twice a day + 1cp200UI once a day) during 24 months (maximum).
  Other Names: PENTO
  Arms: Pentoxifylline and Tocopherol

SUMMARY:
Mandibular osteoradionecrosis, despite its low incidence, remains being the most problematic and irreversible complication after head and neck radiotherapy with no medical treatment to limit or reduce symptoms.

Different clinical trials have shown a significant scientific evidence that the treatment with pentoxifylline + tocopherol achieves a certain effectiveness in the treatment of the tissue fibrosis. This study proposes to use this drugs to determine if there is healing of mandibular osteoradionecrosis and/or a symptomatic improvement as well.

DETAILED DESCRIPTION:
Mandibular osteoradionecrosis which occurs after the use of radiation therapy for the treatment of head and neck cancer remains being the most problematic and irreversible complication despite its low incidence with no medical treatment to limit or reduce symptoms.

Clinical trials conducted to date have shown a significant scientific evidence that the treatment with pentoxifylline + tocopherol achieves a certain effectiveness in the treatment of the tissue fibrosis that have been irradiated based on the properties of this drugs in increased tissue oxygenation and their antioxidant effect.

The aim of this study is to determine if there is a clinical improvement of mandibular osteoradionecrosis using Pentoxifylline in combination with Tocopherol as treatment because, currently, there is no effective treatment to achieve bone healing and/or a symptomatic improvement.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years and under 90 years old.
* Patients who have received radiotherapy after being diagnosed with head and neck cancer and currently are diagnosticated of mandibular osteoradionecrosis (any clinical stage)
* Follow-up for at least a year after the radiation treatment is completed.
* Absence of tumor at the time of recruitment.
* Patients with the capacity to give informed consent

Exclusion Criteria:

* Allergy or hypersensitivity to Pentoxifylline or others xanthines, or to Tocopherol (vitamin E).
* Patients taking oral anticoagulants (acenocoumarol, warfarin).
* Known hemorrhagic/coagulation disorder.
* Vitamin K deficiency due to any cause.
* Use of estrogens oral contraceptives.
* Serious bleeding or extensive retinal hemorrhage.
* Ischaemic heart diseases, including recent Myocardial Infarction.
* Serious cardiac arrhythmia.
* Severe LIVER DISEASE.
* Severe renal failure (creatinine clearance <30 mL/min).
* Hypotension.
* Female patients who are pregnant or lactating
* Any other situation or condition that, in the opinion of the INVESTIGATOR, may interfere with optimal PARTICIPATION in the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Martos-Fernandez, MD, Principal Investigator — Oral and Maxillofacial Surgery (Vall d'Hebrón Hospital)
Locations (1):
- Vall d'Hebrón Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Robard L, Louis MY, Blanchard D, Babin E, Delanian S. Medical treatment of osteoradionecrosis of the mandible by PENTOCLO: preliminary results. Eur Ann Otorhinolaryngol Head Neck Dis. 2014 Dec;131(6):333-338. doi: 10.1016/j.anorl.2013.11.006. Epub 2014 Jun 30. PMID 24993781
- [Background] Delanian S, Chatel C, Porcher R, Depondt J, Lefaix JL. Complete restoration of refractory mandibular osteoradionecrosis by prolonged treatment with a pentoxifylline-tocopherol-clodronate combination (PENTOCLO): a phase II trial. Int J Radiat Oncol Biol Phys. 2011 Jul 1;80(3):832-9. doi: 10.1016/j.ijrobp.2010.03.029. Epub 2010 Jul 16. PMID 20638190
- [Background] Delanian S, Depondt J, Lefaix JL. Major healing of refractory mandible osteoradionecrosis after treatment combining pentoxifylline and tocopherol: a phase II trial. Head Neck. 2005 Feb;27(2):114-23. doi: 10.1002/hed.20121. PMID 15641107

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: No drug treatment
Period: Overall Study
Arm/Group | Pentoxifylline and Tocopherol | Control Group
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline and Tocopherol | Control Group | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (10) | 55 (10) | 56 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 10 | 20
Exposed bone [Mean (Standard Deviation); unit: mm^2] | 10 (10) | 15 (10) | 12.5 (10)

OUTCOME MEASURES:

1. Primary Outcome: Bone and/or Tissue Healing as Measured With the Classification of ORN Stages, Area of Bone Exposed (mm2) and Radiological Findings (OPG).
Description: Clinical healing assessment as measured with the classification of ORN stages, area of bone exposed (mm2) and radiological findings (OPG).
  Intraoral bone exposure is measured in mm2.
Time Frame: From baseline to 1, 3, 6, and 9 months of starting treatment
Population: mean of intraoral bone exposure (measured in mm2) from baseline to 1, 3, 6, 9, 12 and 18 months of starting treatment
Measure: Mean (Full Range); unit: mm2
Groups:
- Control Group: Standard treatment
Arm/Group | Pentoxifylline and Tocopherol | Control Group
Number analyzed (Participants) | 12 | 12
mm2
  1 month of starting treatment | 14 [10 to 18] | 15 [10 to 20]
  3 month of starting treatment | 13 [10 to 16] | 15 [10 to 20]
  6 month of starting treatment | 11.5 [10 to 13] | 15 [10 to 20]
  9 month of starting treatment | 10 [8 to 12] | 15 [10 to 20]

2. Secondary Outcome: Clinical Symptoms Evaluation, Measured Using the LENT-SOMA Scale
Description: Evaluation of symptoms improvement using the LENT-SOMA scale (Late Effect Normal Tissue Task Force / Subjective, Objective, Management, Analytic scale).
  To examine the LENT/SOMA scale prospectively using interviews and questionnaires
  Assessments were made from baseline to 1, 3, 6 and 9 months of starting treatments. The acceptability and feasibility of using the scales was examined using compliance in completion of the questionnaires.
  Maximum score: 36 Minimum score: 0
  Questionnaires have been completed for 24 patients after treatment. Higher values represents worse outcome.
  Scale categories:
  Subjective: pain, nutritional problems, difficulty in mouth openning. Objective: bone exposure, trismus, Management: analgesic treatment, oral treatment, nutrition. Analytic: radiological findings.
Time Frame: From baseline to 1,3, 6, 9 months of starting treatment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Pentoxifylline and Tocopherol | CONTROL
Number analyzed (Participants) | 12 | 12
units on a scale
  1 month of starting treatment | 14.5 [13.2 to 15.8] | 15.5 [14 to 17]
  3 month of starting treatment | 14 [13 to 15] | 15.5 [14 to 17]
  6 month of starting treatment | 14 [13 to 15] | 15.5 [14 to 17]
  9 month of starting treatment | 13.3 [12 to 14.6] | 15.5 [14 to 17]

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Pentoxifylline and Tocopherol | Control Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes